CLINICAL TRIAL: NCT01191541
Title: Treatment of Newly Diagnosed Patients With Acute Promyelocytic Leukemia in Children: Remission Induction With All-transretinoic Acid (ATRA) and Arsenic Trioxide (As2O3). Consolidation With Daunorubicin(DNR)+Ara-c or DNR Alone.
Brief Title: Cytarabine (Ara-C) in Children With Acute Promyelocytic Leukemia (APL)
Acronym: Ara-C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiaofan Zhu (Unknown)
Responsible Party: Sponsor-Investigator, Xiaofan Zhu, chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCAPL2010
Record Dates: First submitted 2010-08-18; First posted 2010-08-31 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Leukemia
Keywords: ara-c; As2O3; pediatric; acute
MeSH Terms: conditions — Leukemia | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DNR+Ara-c(Ara-C group) (Active Comparator): patients in this group were treated with DNR+Ara-C in consolidation
  Interventions: Drug: DNR:; Drug: Ara-c
- DNR(No Ara-C group) (Experimental): patients in this group were treated with DNR alone in consolidation
  Interventions: Drug: DNR:

INTERVENTIONS:
Drug: DNR: — DNR：45mg/m2 d1-3
Drug: Ara-c — DNR+ARA-C：DNR：45mg/m2 d1-3;Ara-C :1g/m2 d1-3
  Arms: DNR+Ara-c(Ara-C group)

SUMMARY:
Several groups, especially the PETHEMA group (in their LPA96 and 99 trials), obtained low relapse rates in newly diagnosed Acute Promyelocytic Leukemia (APL) patients by combining ll-transretinoic acid (ATRA) and anthracyclines without Ara-C, suggesting that avoiding Ara-C in the chemotherapy of APL reduced treatment toxicity without increasing relapses. While the relapse rate for the children with white blood cell(WBC) counts greater than 10×109/L at presentation were higher than those WBC counts less than 10×109/L (31% and 3.5%,respectively) in the LPA96 and 99 trials. A recent adult randomized trial show that avoiding Ara-C leads to an increased risk of relapse in the APL patients with WBC counts less than 10×109/L. The role of the Ara-C remains controversial. And there are very limited data reported on children with APL so far.

DETAILED DESCRIPTION:
Some studies suggest patients with high-risk disease should be treated with intensified doses of anthracycline, or intermediate/ high-dose Ara-C or As2O3 as an early consolidation, so as to decrease the risk of relapse.However, a higher cumulative dose of anthracycline may lead to cardiac toxicity, especially for children. In addition, containing Ara-C will led to more therapy-related toxicity. The benefit to add Ara-C to the schedules is questionable and remains a matter of investigation in children.

ELIGIBILITY:
Inclusion Criteria:

* Acute Promyelocytic Leukemia (APL)

Exclusion Criteria:

* > 14

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofan Zhu, MD, Principal Investigator — Department of Pediatrics, CAMS&PUMC
Locations (2):
- China (2):
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality
  - Department of Pediatrics, Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin, PR China, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ortega JJ, Madero L, Martin G, Verdeguer A, Garcia P, Parody R, Fuster J, Molines A, Novo A, Deben G, Rodriguez A, Conde E, de la Serna J, Allegue MJ, Capote FJ, Gonzalez JD, Bolufer P, Gonzalez M, Sanz MA; PETHEMA Group. Treatment with all-trans retinoic acid and anthracycline monochemotherapy for children with acute promyelocytic leukemia: a multicenter study by the PETHEMA Group. J Clin Oncol. 2005 Oct 20;23(30):7632-40. doi: 10.1200/JCO.2005.01.3359. PMID 16234524
- [Derived] Zhang L, Zou Y, Chen Y, Guo Y, Yang W, Chen X, Wang S, Liu X, Ruan M, Zhang J, Liu T, Liu F, Qi B, An W, Ren Y, Chang L, Zhu X. Role of cytarabine in paediatric acute promyelocytic leukemia treated with the combination of all-trans retinoic acid and arsenic trioxide: a randomized controlled trial. BMC Cancer. 2018 Apr 3;18(1):374. doi: 10.1186/s12885-018-4280-2. PMID 29615003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were those who were less than 14 years old, were newly diagnosed with APL, and had not previously received chemotherapy. Sixty-five patients were included in the study.
Pre-assignment Details: The demonstration of PML-RARA transcripts, was required for inclusion in the analysis.
Groups:
- Daunorubicin(DNR)+Ara-c (Ara-C Group): one group treated with daunorubicin(DNR)+Ara-C in consolidation
- DNR (No Ara-c Group): Only DNR was used in consolidation
Period: All the Patients
Arm/Group | Daunorubicin(DNR)+Ara-c (Ara-C Group) | DNR (No Ara-c Group)
Started | 30 | 35
Completed | 30 | 35
Not Completed | 0 | 0
Period: the Randomized Patients
Arm/Group | Daunorubicin(DNR)+Ara-c (Ara-C Group) | DNR (No Ara-c Group)
Started | 30 | 35
Completed | 30 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DNR+Ara-c: one group treated with DNR+Ara-C
- DNR（ no Ara-C): one group treated with DNR
- Total: Total of all reporting groups
Arm/Group | DNR+Ara-c | DNR（ no Ara-C) | Total
Number analyzed (Participants) | 30 | 35 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 35 | 65
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 8 [2 to 13] | 7 [2 to 14] | 8 [2 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 20 | 22 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants] — Eligible patients were less than 14 years of age with newly diagnosed APL without chemotherapy used before. Molecular diagnosis was not required for enrollment, but subsequent molecular confirmation by demonstration of promyelocytic leukemia(PML)-retinoic acid receptor alpha(RARA)（PML-RARA） transcripts was required for inclusion in the analysis. A genetic diagnosis could be established by detection of the PML-RARA fusion gene by means of polymerase-chain-reaction (PCR) assay Population: Between May 2010 and December 2016, 65 consecutive patients with genetically confirmed newly diagnosed APL patients (≤14years) were admitted in our hospital.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 30 | 35 | 65
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 30 | 35 | 65
white blood cell count [Median (Full Range); unit: cells x 10^9/L] | 4.23 [0.99 to 130] | 5.47 [0.82 to 202.4] | 4.71 [0.82 to 202.4]
Haemoglobin [Median (Full Range); unit: g/L] | 78 [44 to 124] | 81.0 [49 to 127] | 78 [44 to 124]
Platelet count [Median (Full Range); unit: cells x 10^9/L] | 24.5 [2 to 125] | 32.0 [6 to 130] | 30.5 [2 to 130]

OUTCOME MEASURES:

1. Primary Outcome: the Overall Survival of APL Patients Treated With Retinoic Acid Receptor Alpha (ATRA) and Arsenic Trioxide (ATO) Based Trial
Description: We assessed the OS of APL patients when ATRA and ATO were used. The overall survival (OS) durations was calculated from the date of diagnosis to last follow-up or death.
Time Frame: two years
Population: There were 65 patients included in our study, including 35 in the DNR group and 30 in the DNR+Ara-C group.
Measure: Number; unit: participants
Groups:
- DNR Group: the patients in this group were treated with DNR alone in consolidation
- DNR+Ara-C Group: the patients in this group were treated with DNR +Ara-C in consolidation
Arm/Group | DNR Group | DNR+Ara-C Group
Number analyzed (Participants) | 35 | 30
participants
  relapse | 1 | 0
  died | 0 | 0
Statistical Analysis 1: Comparison: DNR Group vs DNR+Ara-C Group; The characteristics of all of the included patients were summarized using cross-tabulations (for categorical variables) and quantiles. Nonparametric tests were used to analyse comparisons between groups .EFS、disease-free survival (DFS) and OS were estimated using the Kaplan -Meier method, and log-rank tests were used. All P values were two-sided, and those with values of 0.05 or less were considered to be statistically significant; Test type: Non-Inferiority — The primary objective was to demonstrate the noninferiority of DNR alone to DNR+ARA-C in the rate of DFS at 2 years. Assuming a 95% rate of DFS in the two groups, a margin of -15% , 5% type 1 error, 80% power, 30 evaluable patients per group were required to draw a noninferiority conclusion; p < 0.05, Log Rank — the p-value is not adjusted

2. Primary Outcome: the Event-free Survival (EFS） of APL Patients Treated With Retinoic Acid Receptor Alpha (ATRA) and Arsenic Trioxide (ATO) Based Trial
Description: We assessed the EFS of APL patients treated with retinoic acid receptor alpha (ATRA) and Arsenic Trioxide (ATO) based trial. Event-free survival (EFS) was defined as time from diagnosis to last follow-up or an event (relapse or death).
Time Frame: 2 years
Population: There were 65 patients included in our study, including 35 in the DNR group and 30 in the DNR+Ara-C group.
Measure: Number; unit: participants
Arm/Group | DNR+Ara-c(Ara-C Group) | DNR(No Ara-C Group)
Number analyzed (Participants) | 30 | 35
participants
  relapse | 0 | 1
  die | 0 | 0

3. Secondary Outcome: Number of Participants With Side Effects
Description: Also, we compared the side effect and outcome between the two groups.To assessed whether Ara-C could be omitted when ATO and ATRA were used.
Time Frame: three years
Population: There were 66 patients included in our study. One patient gave up treatment due to the economic reasons. Then the number of the patients were 65, including 35 in the DNR group and 30 in the DNR+Ara-C group.
Measure: Count of Participants; unit: Participants
Groups:
- DNR+Ara-c (Ara-C Group): one group treated with DNR+Ara-C in consolidation
Arm/Group | DNR+Ara-c (Ara-C Group) | DNR (No Ara-c Group)
Number analyzed (Participants) | 30 | 35
Participants
  sepsis | 5 | 1
  platelet transfusion | 26 | 0
  red blood cell transfusion | 7 | 7
  relapse | 0 | 1

ADVERSE EVENTS:
Time Frame: Between May 2010 and December 2016, 65 consecutive paediatric (≤14years old) patients who were genetically confirmed with a new diagnosis of APL were admitted in our hospital.The follow-up of the patients was updated on Jan 2017 and included a median of 32 months (range, 1 to 79). The adverse event data were collected from the patient enrolled in our trials.The median period of time were 32 months (range, 1 to 79).
Description: All adverse events described were founded during the course of induction therapy.
Groups:
- All the Patients at Presentation: Between May 2010 and December 2016, 65 consecutive paediatric (≤14 years of age) patients who were genetically confirmed with a new diagnosis of APL were admitted in our hospital.
- the Adverse Events Associated With ATRA; the Adverse Events Associated With ATO: There were 65 patients were treated with ATRA and ATO in induction.
- Consolidation: IDA: There were 65 patients were treated with IDA in consolidation. .
- Consolidation: ATO: There were 65 patients were treated with ATO in consolidation.
- Consolidation: DNR (No Ara-c Group): There were 35 patients were treated with DNR in consolidation.
- Consolidation: DNR+Ara-c (Ara-C Group): There were 30 patients were treated with DNR+ARA-C in consolidation.
- Maintenance: ATRA+MTX+6-MP: There were 65 patients were treated with maintenance.
Arm/Group | All the Patients at Presentation | the Adverse Events Associated With ATRA | the Adverse Events Associated With ATO | Consolidation: IDA | Consolidation: ATO | Consolidation: DNR (No Ara-c Group) | Consolidation: DNR+Ara-c (Ara-C Group) | Maintenance: ATRA+MTX+6-MP
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65 | 0/65 | 0/65 | 0/65 | 0/35 | 0/30 | 0/65
Serious Adverse Events (participants affected / at risk) | 12/65 | 2/65 | 1/65 | 0/65 | 0/65 | 0/35 | 0/30 | 0/65
Other Adverse Events (participants affected / at risk) | 0/65 | 55/65 | 21/65 | 3/65 | 0/65 | 0/35 | 0/30 | 0/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | All the Patients at Presentation (N=65) | the Adverse Events Associated With ATRA (N=65) | the Adverse Events Associated With ATO (N=65) | Consolidation: IDA (N=65) | Consolidation: ATO (N=65) | Consolidation: DNR (No Ara-c Group) (N=35) | Consolidation: DNR+Ara-c (Ara-C Group) (N=30) | Maintenance: ATRA+MTX+6-MP (N=65)
intracranial bleeding (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/30 (0) | 0 (0) | 0 (0)
intraocular bleeding (Eye disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
mild partial splenic embolization (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
retinoic acid syndrome (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cardiac arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All the Patients at Presentation (N=65) | the Adverse Events Associated With ATRA (N=65) | the Adverse Events Associated With ATO (N=65) | Consolidation: IDA (N=65) | Consolidation: ATO (N=65) | Consolidation: DNR (No Ara-c Group) (N=35) | Consolidation: DNR+Ara-c (Ara-C Group) (N=30) | Maintenance: ATRA+MTX+6-MP (N=65)
extremity oedema (General disorders) | 0 (0) | 0 (0) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
skin pigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
bone ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
asymptomatic QTc prolongation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
headache (General disorders) | 0 (0) | 24 (24) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
retinoic acid syndrome (Blood and lymphatic system disorders) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2010-08-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT01191541/Prot_000.pdf
  • Statistical Analysis Plan (2010-08-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT01191541/SAP_001.pdf